CLINICAL TRIAL: NCT00432042
Title: An Open, Randomised, Comparative, Multicentre Study of the Immunogenicity and Safety of Concomitant Versus Separate Administration of a Combined Measles, Mumps, Rubella and Varicella Live Vaccine (ProQuad®) and a Booster Dose of Infanrix® Hexa in Healthy Children 12 to 23 Months of Age
Brief Title: Immunogenicity and Safety Study of Proquad® and Infanrix® Hexa When Administered Concomitantly (V221-035)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V221-035; X06-MMRV-302 (Other: Sanofi Pasteur MSD Protocol Number); 2006-004129-27 (EudraCT Number)
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-02

CONDITIONS: Varicella; Measles; Mumps; Rubella; Diphtheria; Tetanus; Pertussis; Poliomyelitis; Hepatitis B; Haemophilus Infections
Keywords: Mumps and Rubella; Haemophilus influenzae type b (Infanrix® hexa)
MeSH Terms: conditions — Chickenpox; Measles; Mumps; Rubella; Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Hepatitis B; Haemophilus Infections | interventions — measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ProQuad® + Infanrix® hexa (Experimental): Pediatric (12 to 23 months of age) participants received ProQuad® and Infanrix® hexa (booster dose) concomitantly on Visit 1 (Day 0). Blood samples were taken on Visit 1 and Visit 2 (Day 42).
  Interventions: Biological: ProQuad®; Biological: Infanrix® hexa
- ProQuad® (Active Comparator): Pediatric (12 to 23 months of age) participants received ProQuad® on Visit 1 (Day 0). Blood samples were taken on Visit 1 and Visit 2 (Day 42).
  Interventions: Biological: ProQuad®
- Infanrix® hexa (Active Comparator): Pediatric (12 to 23 months of age) participants received Infanrix® hexa (booster dose) on Visit 1 (Day 0). Blood samples were taken on Visit 1 and Visit 2 (Day 42).
  Interventions: Biological: Infanrix® hexa

INTERVENTIONS:
Biological: ProQuad® — Participants received a 0.5 mL subcutaneous injection of ProQuad® containing the following live attenuated virus strains: measles virus Enders' Edmonston strain (≥3.00 log10 50% cell culture infectious dose [CCID]50), mumps virus Jeryl Lynn™ (Level B) strain (≥4.30 log10 CCID50), rubella virus Wistar RA 27/3 strain (≥3.00 log10 CCID50), and varicella virus Oka/Merck strain (≥3.99 log10 plaque-forming units [PFU]).
  Arms: ProQuad®; ProQuad® + Infanrix® hexa
Biological: Infanrix® hexa — Participants received a 0.5 mL intramuscular injection of Infanrix® hexa containing the following: diphtheria toxoid (≥30 IU), tetanus toxoid (≥40 IU), 3-component acellular pertussis (pertussis taxoid, filamentous haemagglutinin, and pertactin) (25 ug), Hepatitis B surface antigen recombinant (S protein) (10 ug), inactivated poliovirus types 1-3 (type 1: 40 D-antigen units; type 2: 8 D-antigen units; type 3: 32 D-antigen units), and Haemophilus influenzae type B (Hib) polysaccharide conjugate to tetanus toxoid (20-40 ug).
  Arms: Infanrix® hexa; ProQuad® + Infanrix® hexa

SUMMARY:
Primary Objective:

* To demonstrate that ProQuad® can be administered concomitantly with a booster dose of Infanrix® hexa to healthy children 12 to 23 months of age without impairing either the antibody response rates to measles, mumps, rubella, varicella, hepatitis B and Haemophilus influenzae type b; or to the 3 pertussis antibody titres measured at 42 days following vaccination.

Secondary Objectives:

* To describe the antibody titres and the antibody response rates to measles, mumps, rubella, varicella, diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis and Haemophilus influenzae type b as measured at 42 days following vaccination by an Infanrix® hexa primary series schedule and all data are pooled.
* To evaluate the safety profile of ProQuad® when administered concomitantly with a booster dose of Infanrix® hexa by an Infanrix® hexa primary series schedule and all data are pooled.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants of either gender
* Aged 12 to 23 months
* No clinical history of measles, mumps, rubella, varicella and zoster
* For Italy: Primary vaccination with the combined diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis and Haemophilus influenzae type b vaccine Infanrix® hexa as a 2-dose schedule, with receipt of the second dose ≥ 6 months prior to inclusion
* For Germany: Primary vaccination with the combined diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis and Haemophilus influenzae type b vaccine Infanrix® hexa as a 3-dose schedule, with receipt of the third dose ≥ 6 months prior to inclusion
* Consent form signed by parent(s) according to local regulations or by the legal representative properly informed about the study
* Parent(s)/legal representative able to understand the protocol requirements and to fill in the Diary Card.

Exclusion Criteria:

* Prior receipt of measles, mumps, rubella and/or varicella vaccine either alone or in any combination
* Any recent (<= 30 days) exposure to measles, mumps, rubella, varicella and/or zoster
* Receipt of any other diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis and/or Haemophilus influenzae type b containing vaccine (either alone or in any combination) than Infanrix® hexa
* Any recent (<= 3 days) history of febrile illness
* Any severe chronic disease
* Active untreated tuberculosis
* Known personal history of encephalopathy, seizure disorder or progressive, evolving or unstable neurological condition
* Any known blood dyscrasia, leukemia, lymphomas of any type, or other malignant neoplasms affecting the haematopoietic or lymphatic systems
* Any severe thrombocytopenia or any other coagulation disorder that would contraindicate intramuscular injection
* Prior known sensitivity/allergy to any component of the vaccines including neomycin, sorbitol or gelatin
* Any immune impairment or humoral/cellular deficiency, neoplastic disease or depressed immunity
* Any recent (<= 2 days) tuberculin test or scheduled tuberculin test through Visit 2
* Any previous (<= 150 days) receipt of immune serum globulin or any blood-derived products or scheduled to be administered through Visit 2
* Any recent (<= 30 days) receipt of an inactivated or a live non-study vaccine or scheduled non-study vaccination through Visit 2
* Any medical condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives
* Any recent (≤30 days) participation or scheduled participation in any other clinical trial through Visit 2

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 955 (Actual)
Dates: Start 2007-01-12 (Actual); Primary Completion 2008-03-27 (Actual); Study Completion 2008-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Fiquet, MD, Study Director — SPMSD
Locations (50):
- Germany (44):
  - Alsfeld
  - Bad Saulgau
  - Bad Säckingen
  - Bad Sobernheim
  - Berlin
  - Bielefeld
  - Birkenfeld
  - Bramsche
  - Bretten
  - Brunsbüttel
  - Datteln
  - Detmold
  - Espelkamp
  - Ettenheim
  - Friedrichshafen
  - Gerolstein
  - Gifhorn
  - Gütersloh
  - Hamburg
  - Heilbronn
  - Herbolzheim
  - Karlsruhe
  - Kehl
  - Koblenz
  - Lauffen am Neckar
  - Mannheim
  - Marbach
  - Mönchengladbach
  - München
  - Neustadt A.d. Aisch
  - Nidderau
  - Oberhausen
  - Oberkirch
  - Offenburg
  - Pegnitz
  - Rodorf
  - Schwäbisch Hall
  - Schwieberdingen
  - Traunreut
  - Veitshöchheim
  - Wanzleben
  - Welzheim
  - Wildeshausen
  - Zwiesel
- Italy (6):
  - Chiavari
  - Ferrara
  - Latisana
  - Ragusa
  - Sassari
  - Taranto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deichmann KA, Ferrera G, Tran C, Thomas S, Eymin C, Baudin M. Immunogenicity and safety of a combined measles, mumps, rubella and varicella live vaccine (ProQuad (R)) administered concomitantly with a booster dose of a hexavalent vaccine in 12-23-month-old infants. Vaccine. 2015 May 11;33(20):2379-86. doi: 10.1016/j.vaccine.2015.02.070. Epub 2015 Mar 9. PMID 25765966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 963 participants were screened at study centers in Italy and Germany.
Groups:
- Arm 1: ProQuad® + Infanrix® Hexa: Pediatric (12 to 23 months of age) participants received ProQuad® and Infanrix® hexa (booster dose) concomitantly on Visit 1 (Day 0). Blood samples were taken on Visit 1 and Visit 2 (Day 42).
- Arm 2: ProQuad®: Pediatric (12 to 23 months of age) participants received ProQuad® on Visit 1 (Day 0). Blood samples were taken on Visit 1 and Visit 2 (Day 42).
- Arm 3: Infanrix® Hexa: Pediatric (12 to 23 months of age) participants received Infanrix® hexa (booster dose) on Visit 1 (Day 0). Blood samples were taken on Visit 1 and Visit 2 (Day 42).
Period: Overall Study
Arm/Group | Arm 1: ProQuad® + Infanrix® Hexa | Arm 2: ProQuad® | Arm 3: Infanrix® Hexa
Started | 479 (Number randomized.) | 235 (Number randomized.) | 241 (Number randomized.)
Vaccinated | 477 | 235 | 240
Completed | 472 | 234 | 239
Not Completed | 7 | 1 | 2
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Lost to Follow-up | 5 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: ProQuad® + Infanrix® Hexa | Arm 2: ProQuad® | Arm 3: Infanrix® Hexa | Total
Number analyzed (Participants) | 479 | 235 | 241 | 955
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.6 (1.9) | 13.4 (1.5) | 13.5 (1.7) | 13.5 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 112 | 114 | 448
  Male | 257 | 123 | 127 | 507

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting Antibody Response Rate Criteria to Measles, Mumps, Rubella, and Varicella
Description: The percentage of participants with seronegative baseline values who met antibody response criteria in Arm 1: ProQuad® + Infanrix® hexa and Arm 2: ProQuad® was determined. Post-vaccination antibody response and baseline seronegativity criteria were as follows: measles antibody titre ≥255 mIU/mL in participants with baseline titre <255 mIU/mL; mumps antibody titre ≥10 ELISA Ab units/mL in participants with baseline titre <10 ELISA Ab units mL; rubella antibody titre ≥10 IU/mL in participants with baseline titre <10 IU/mL; varicella antibody titre ≥5 gpELISA units/mL in participants with baseline titre <1.25 gpELISA units/mL. Measles, mumps and rubella antibody levels were determined using enzyme-linked immunosorbent assay (ELISA) and varicella antibody levels were determined with glycoprotein-based ELISA (gpELISA).
Time Frame: Day 42
Population: Participants in Arm 1 and Arm 2 who were initially seronegative to measles, mumps, rubella, or varicella; had post-vaccination serology results; and who did not have protocol violations that may have interfered with immunogenicity results were included. As analysis of Arm 3 was not planned it was not included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1: ProQuad® + Infanrix® Hexa | Arm 2: ProQuad®
Number analyzed (Participants) | 431 | 215
Percentage of Participants
  Measles: number analyzed (Participants) | 421 | 215
  Measles | 97.4 [95.4 to 98.7] | 96.3 [92.8 to 98.4]
  Mumps: number analyzed (Participants) | 427 | 212
  Mumps | 96.7 [94.6 to 98.2] | 98.6 [95.9 to 99.7]
  Rubella | 97.9 [96.1 to 99.0] | 99.1 [96.7 to 99.9]
  Varicella: number analyzed (Participants) | 394 | 205
  Varicella | 97.7 [95.7 to 99.0] | 95.1 [91.2 to 97.6]
Statistical Analysis 1: Comparison: Arm 1: ProQuad® + Infanrix® Hexa vs Arm 2: ProQuad®; Test type: Non-Inferiority or Equivalence — Measles difference; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [-1.62 to 4.82] — Non-inferiority was declared when the lower bound of the two-sided 95% CI of the difference is > -10%
Statistical Analysis 2: Comparison: Arm 1: ProQuad® + Infanrix® Hexa vs Arm 2: ProQuad®; Test type: Non-Inferiority or Equivalence — Mumps difference; Mean Difference (Final Values) = -1.83, 95% CI 2-sided [-4.21 to 1.10] — Non-inferiority was declared when the lower bound of the two-sided 95% CI of the difference is > -10%
Statistical Analysis 3: Comparison: Arm 1: ProQuad® + Infanrix® Hexa vs Arm 2: ProQuad®; Test type: Non-Inferiority or Equivalence — Rubella difference; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-3.19 to 1.35] — Non-inferiority was declared when the lower bound of the two-sided 95% CI of the difference is > -10%
Statistical Analysis 4: Comparison: Arm 1: ProQuad® + Infanrix® Hexa vs Arm 2: ProQuad®; Test type: Non-Inferiority or Equivalence — Varicella difference; Mean Difference (Final Values) = 2.53, 95% CI 2-sided [-0.41 to 6.58] — Non-inferiority was declared when the lower bound of the two-sided 95% CI of the difference is > -10%

2. Primary Outcome: Percentage of Participants Meeting Post-vaccination Antibody Response Rates to Hepatitis B and Haemophilus Influenzae Type B
Description: The percentage of participants with seronegative baseline values who met antibody response criteria in Arm 1: ProQuad® + Infanrix® hexa and Arm 3: Infanrix® hexa was determined. Post-vaccination antibody response and baseline seronegativity criteria were as follows: Hepatitis B antibody titre ≥10 IU/mL and Haemophilus Influenzae Type b antibody titre ≥1 ug/mL. Hepatitis B antibody levels were determined using anti-HBs ORTHO ECi Immunodiagnostic Assay. Haemophilus Influenzae Type b antibody (anti-polyribosylribitol phosphate [PRP]) levels were determined with radioimmunoassay (RIA) or with enzyme immunoassay (EIA).
Time Frame: Day 42
Population: Participants in Arm 1 and Arm 3 who had post-vaccination serology results and who did not have protocol violations that may have interfered with immunogenicity results were included. As analysis of Arm 2 was not planned it was not included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ProQuad® + Infanrix® Hexa | Arm 3: Infanrix® Hexa
Number analyzed (Participants) | 411 | 215
Percentage of participants
  Hepatitis B | 99.5 [98.3 to 99.9] | 98.1 [95.3 to 99.5]
  Haemophilus Influenzae Type B: number analyzed (Participants) | 387 | 211
  Haemophilus Influenzae Type B | 98.2 [96.3 to 99.3] | 95.3 [91.5 to 97.7]
Statistical Analysis 1: Comparison: Arm 1: ProQuad® + Infanrix® Hexa vs Arm 3: Infanrix® Hexa; Test type: Non-Inferiority or Equivalence — Hepatitis B difference; Mean Difference (Final Values) = 1.36, 95% CI 2-sided [-0.29 to 4.24] — Non-inferiority was declared when the lower bound of the two-sided 95% CI of the difference is > -5%
Statistical Analysis 2: Comparison: Arm 1: ProQuad® + Infanrix® Hexa vs Arm 3: Infanrix® Hexa; Test type: Non-Inferiority or Equivalence — Haemophilus Influenza type B difference; Mean Difference (Final Values) = 2.97, 95% CI 2-sided [-0.17 to 6.89] — Non-inferiority was declared when the lower bound of the two-sided 95% CI of the difference is > -5%

3. Primary Outcome: Post-vaccination Geometric Mean Titres (GMT) to Pertussis
Description: The GMT to pertussis were compared in Arm1: ProQuad® + Infanrix® hexa and Arm 3: Infanrix® hexa. Anti-pertussis toxin (anti-PT), anti-filamentous hemagglutinin (anti-FHA), and anti-pertactin (anti-PRN) were determined using ELISA on solid phase based on sandwich principle.
Time Frame: Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: GMT (IU/mL)
Arm/Group | Arm 1: ProQuad® + Infanrix® Hexa | Arm 3: Infanrix® Hexa
Number analyzed (Participants) | 386 | 211
GMT (IU/mL)
  Anti-PT GMT: number analyzed (Participants) | 379 | 211
  Anti-PT GMT | 132.6 [123.8 to 142.0] | 139.1 [126.7 to 152.8]
  Anti-FHA GMT | 210.9 [195.7 to 227.2] | 189.9 [170.2 to 211.8]
  Anti-PRN GMT: number analyzed (Participants) | 385 | 211
  Anti-PRN GMT | 310.0 [282.2 to 340.7] | 259.7 [226.3 to 298.1]
Statistical Analysis 1: Comparison: Arm 1: ProQuad® + Infanrix® Hexa; Test type: Non-Inferiority or Equivalence — Anti-PT difference; GMT ratio = 0.97, 95% CI 2-sided [0.88 to 1.08] — Non-inferiority was declared when the lower bound of the two-sided 95% CI of the difference is > -5%
Statistical Analysis 2: Comparison: Arm 1: ProQuad® + Infanrix® Hexa; Test type: Non-Inferiority or Equivalence — Anti-FHA difference; GMT ratio = 1.09, 95% CI 2-sided [0.98 to 1.23] — Non-inferiority was declared when the lower bound of the two-sided 95% CI of the difference is > -5%
Statistical Analysis 3: Comparison: Arm 1: ProQuad® + Infanrix® Hexa vs Arm 3: Infanrix® Hexa; Test type: Non-Inferiority or Equivalence — Anti-PRN difference; GMT ratio = 1.18, 95% CI 2-sided [1.03 to 1.36] — Non-inferiority was declared when the lower bound of the two-sided 95% CI of the difference is > -5%

ADVERSE EVENTS:
Time Frame: Up to Day 42
Description: All participants who received at least one dose of study vaccine and who have safety follow-up data are included.
Arm/Group | Arm 1: ProQuad® + Infanrix® Hexa | Arm 2: ProQuad® | Infanrix® Hexa
Serious Adverse Events (participants affected / at risk) | 7/474 | 6/234 | 4/239
Other Adverse Events (participants affected / at risk) | 409/474 | 134/234 | 184/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: ProQuad® + Infanrix® Hexa (N=474) | Arm 2: ProQuad® (N=234) | Infanrix® Hexa (N=239)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Electric shock (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: ProQuad® + Infanrix® Hexa (N=474) | Arm 2: ProQuad® (N=234) | Infanrix® Hexa (N=239)
Diarrhoea (Gastrointestinal disorders) | 22 (23) | 14 (14) | 14 (14)
Vomiting (Gastrointestinal disorders) | 14 (15) | 2 (2) | 14 (15)
Injection site erythema (General disorders) | 274 (338) | 31 (31) | 126 (131)
Injection site pain (General disorders) | 198 (285) | 33 (33) | 84 (84)
Injection site swelling (General disorders) | 203 (235) | 7 (7) | 93 (93)
Pyrexia (General disorders) | 184 (263) | 80 (104) | 68 (91)
Bronchitis (Infections and infestations) | 27 (28) | 12 (12) | 12 (12)
Nasopharyngitis (Infections and infestations) | 48 (50) | 14 (16) | 18 (18)
Rhinitis (Infections and infestations) | 27 (28) | 20 (23) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (32) | 13 (15) | 11 (11)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 33 (36) | 16 (16) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sanofi Pasteur MSD shall have sixty days to review these documents and may refuse to give its consent in part or whole for confidential reasons (including but not limited to intellectual property rights, whether patentable or not).